CLINICAL TRIAL: NCT05429515
Title: Effect of HFR-SUPRA in the Treatment of Multiple Myeloma-related Acute Kidney Injury: a Prospective Cohort Study
Brief Title: Effect of HFR-SUPRA in the Treatment of Multiple Myeloma-related Acute Kidney Injury
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Bellco Hoxen Medical (Shanghai) Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HFR_MM
Record Dates: First submitted 2022-06-19; First posted 2022-06-23 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2022-04

CONDITIONS: Multiple Myeloma; Acute Kidney Injury; Hemodiafiltration With Ultrafiltrate Regeneration (HFR)
MeSH Terms: conditions — Multiple Myeloma; Acute Kidney Injury | interventions — Hemodiafiltration; Renal Dialysis; Drug Therapy

STUDY DESIGN:
Intervention Model Description: Patients are divided into two groups: (1) chemotherapy combined with HFR-SUPRA (2) chemotherapy combined with hemodialysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFR-SUPRA (Experimental): haemodiafiltration with ultrafiltrate regeneration by adsorption on resin (HFR-SUPRA) combined with chemotherapy. HFR-SUPRA everyday for 3 days, then 3 times per week.
  Interventions: Procedure: HFR-SUPRA; Drug: Chemotherapy
- Hemodialysis (Active Comparator): hemodialysis combined with chemotherapy. Hemodialysis everyday for 3 days, then 3 times per week.
  Interventions: Procedure: hemodialysis; Drug: Chemotherapy

INTERVENTIONS:
Procedure: HFR-SUPRA — HFR-SUPRA everyday for 3 days, then 3 times/week until patients do not require dialysis.
  Other Names: haemodiafiltration with ultrafiltrate regeneration by adsorption on resin
  Arms: HFR-SUPRA
Procedure: hemodialysis — hemodialysis everyday for 3 days, then 3 times/week until patients do not require dialysis.
  Arms: Hemodialysis
Drug: Chemotherapy — chemotherapy protocol will be made by hematologists.

SUMMARY:
In patients with multiple myeloma-related acute kidney injury, compare the renal outcome of chemotherapy combined with HFR-SUPRA to chemotherapy combined with hemodialysis.

DETAILED DESCRIPTION:
In patients with multiple myeloma-related severe acute kidney injury, compare the renal outcome between patients receiving HFR-SUPRA and patients receiving hemodialysis. Both groups of patients receive chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* new onset of multiple myeloma
* acute kidney injury with eGFR < 15 ml/min/1.73m2 and need hemodialysis
* biopsy-proven cast nephropathy or clinical diagnosis of cast nephropathy based on exclusion of other causes of acute kidney injury including post-renal obstruction, hypercalcaemia, amyloidosis, light-chain deposition disease, contrast media and drug nephropathy
* serum light chain > 500 mg/L

Exclusion Criteria:

* chronic kidney disease stage 3 to 5 (eGFR< 60 ml/min/1.73m2 for at least 3 months)
* haemodynamics unstability
* active bleeding
* cardiovascular and cerebrovascular events in the last month
* other malignant tumor
* conditions not suitable to participate in the study, such as bad compliance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2032-07-01 (Estimated); Study Completion 2032-12-01 (Estimated)

PRIMARY OUTCOMES:
independence from dialysis at 90 days from allocation to groups | 90 days after allocation to groups
  independence from dialysis at 90 days from allocation to groups

SECONDARY OUTCOMES:
independence from dialysis at 6 months from allocation to groups | 6 months after allocation to groups
  independence from dialysis at 6 months from allocation to groups
complete renal recovery at 90 days from allocation to groups | 90 days after allocation to groups
  serum creatinine elevation≤ 0.2 mg/dl from baseline or serum creatinine ≤ 1.2 mg/dl if baseline level is unknown
decline of free light chain at 21 days from allocation to groups | 21 days after allocation to groups
  decline of free light chain from baseline level
hematological remission at 90 days from allocation to groups | 90 days after allocation to groups
  hematological remission at 90 days from allocation to groups
hematological remission at 6 months from allocation to groups | 6 months after allocation to groups
  hematological remission at 6 months from allocation to groups
time to independence from dialysis | from allocation to groups to the last time of Hemodialysis or HFR-SUPRA
  time to independence from dialysis
survival at 12 months | 12 months after allocation to groups
  survival at 12 months
adverse events | within the 3 months after allocation to groups
  adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Qin, MD, Principal Investigator — Peking Union Medical College Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajkumar SV, Dimopoulos MA, Palumbo A, Blade J, Merlini G, Mateos MV, Kumar S, Hillengass J, Kastritis E, Richardson P, Landgren O, Paiva B, Dispenzieri A, Weiss B, LeLeu X, Zweegman S, Lonial S, Rosinol L, Zamagni E, Jagannath S, Sezer O, Kristinsson SY, Caers J, Usmani SZ, Lahuerta JJ, Johnsen HE, Beksac M, Cavo M, Goldschmidt H, Terpos E, Kyle RA, Anderson KC, Durie BG, Miguel JF. International Myeloma Working Group updated criteria for the diagnosis of multiple myeloma. Lancet Oncol. 2014 Nov;15(12):e538-48. doi: 10.1016/S1470-2045(14)70442-5. Epub 2014 Oct 26. PMID 25439696
- [Background] Dimopoulos MA, Delimpasi S, Katodritou E, Vassou A, Kyrtsonis MC, Repousis P, Kartasis Z, Parcharidou A, Michael M, Michalis E, Gika D, Symeonidis A, Pouli A, Konstantopoulos K, Terpos E, Kastritis E. Significant improvement in the survival of patients with multiple myeloma presenting with severe renal impairment after the introduction of novel agents. Ann Oncol. 2014 Jan;25(1):195-200. doi: 10.1093/annonc/mdt483. PMID 24356630
- [Background] Sanders PW. Mechanisms of light chain injury along the tubular nephron. J Am Soc Nephrol. 2012 Nov;23(11):1777-81. doi: 10.1681/ASN.2012040388. Epub 2012 Sep 20. PMID 22997259
- [Background] Hutchison CA, Batuman V, Behrens J, Bridoux F, Sirac C, Dispenzieri A, Herrera GA, Lachmann H, Sanders PW; International Kidney and Monoclonal Gammopathy Research Group. The pathogenesis and diagnosis of acute kidney injury in multiple myeloma. Nat Rev Nephrol. 2011 Nov 1;8(1):43-51. doi: 10.1038/nrneph.2011.168. PMID 22045243
- [Background] Hutchison CA, Cockwell P, Stringer S, Bradwell A, Cook M, Gertz MA, Dispenzieri A, Winters JL, Kumar S, Rajkumar SV, Kyle RA, Leung N. Early reduction of serum-free light chains associates with renal recovery in myeloma kidney. J Am Soc Nephrol. 2011 Jun;22(6):1129-36. doi: 10.1681/ASN.2010080857. Epub 2011 Apr 21. PMID 21511832
- [Background] Heyne N, Denecke B, Guthoff M, Oehrlein K, Kanz L, Haring HU, Weisel KC. Extracorporeal light chain elimination: high cut-off (HCO) hemodialysis parallel to chemotherapy allows for a high proportion of renal recovery in multiple myeloma patients with dialysis-dependent acute kidney injury. Ann Hematol. 2012 May;91(5):729-735. doi: 10.1007/s00277-011-1383-0. Epub 2011 Dec 15. PMID 22170517
- [Background] Bridoux F, Carron PL, Pegourie B, Alamartine E, Augeul-Meunier K, Karras A, Joly B, Peraldi MN, Arnulf B, Vigneau C, Lamy T, Wynckel A, Kolb B, Royer B, Rabot N, Benboubker L, Combe C, Jaccard A, Moulin B, Knebelmann B, Chevret S, Fermand JP; MYRE Study Group. Effect of High-Cutoff Hemodialysis vs Conventional Hemodialysis on Hemodialysis Independence Among Patients With Myeloma Cast Nephropathy: A Randomized Clinical Trial. JAMA. 2017 Dec 5;318(21):2099-2110. doi: 10.1001/jama.2017.17924. PMID 29209721
- [Background] Hutchison CA, Cockwell P, Moroz V, Bradwell AR, Fifer L, Gillmore JD, Jesky MD, Storr M, Wessels J, Winearls CG, Weisel K, Heyne N, Cook M. High cutoff versus high-flux haemodialysis for myeloma cast nephropathy in patients receiving bortezomib-based chemotherapy (EuLITE): a phase 2 randomised controlled trial. Lancet Haematol. 2019 Apr;6(4):e217-e228. doi: 10.1016/S2352-3026(19)30014-6. Epub 2019 Mar 11. PMID 30872075
- [Background] Pendon-Ruiz de Mier MV, Alvarez-Lara MA, Ojeda-Lopez R, Martin-Malo A, Carracedo J, Caballero-Villarraso J, Alonso C, Aljama P. Effectiveness of haemodiafiltration with ultrafiltrate regeneration in the reduction of light chains in multiple myeloma with renal failure. Nefrologia. 2013 Nov 13;33(6):788-96. doi: 10.3265/Nefrologia.pre2013.Sep.12176. English, Spanish. PMID 24241366
- [Background] Pendon-Ruiz de Mier MV, Ojeda R, Alvarez-Lara MA, Navas A, Alonso C, Caballero-Villarraso J, Aljama P, Alvarez MA, Soriano S, Rodriguez M, Martin-Malo A. Hemodiafiltration with ultrafiltrate regeneration reduces free light chains without albumin loss in multiple myeloma patients. BMC Nephrol. 2020 Jun 15;21(1):227. doi: 10.1186/s12882-020-01885-8. PMID 32539688
- [Background] Mene P, Giammarioli E, Fofi C, Antolino G, Verde G, Tafuri A, Punzo G, Festuccia F. Serum Free Light Chains Removal by HFR Hemodiafiltration in Patients with Multiple Myeloma and Acute Kidney Injury: a Case Series. Kidney Blood Press Res. 2018;43(4):1263-1272. doi: 10.1159/000492408. Epub 2018 Aug 3. PMID 30078004